CLINICAL TRIAL: NCT02327078
Title: A Phase 1/2 Study of the Safety, Tolerability, and Efficacy of Epacadostat Administered in Combination With Nivolumab in Select Advanced Cancers (ECHO-204)
Brief Title: A Study of the Safety, Tolerability, and Efficacy of Epacadostat Administered in Combination With Nivolumab in Select Advanced Cancers (ECHO-204)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 24360-204 / ECHO-204; 2016-002423-29 (EudraCT Number)
Record Dates: First submitted 2014-12-01; First posted 2014-12-30 (Estimated); Results first posted 2023-04-26 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: B-cell Malignancies; Colorectal Cancer (CRC); Head and Neck Cancer; Lung Cancer; Lymphoma; Melanoma; Ovarian Cancer; Glioblastoma
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Lymphoma; Melanoma; Ovarian Neoplasms; Glioblastoma | interventions — Nivolumab; epacadostat; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Phase 1 Part 1 Epacadostat 25mg BID +Nivolumab (Experimental): Epacadostat 25mg oral twice daily (BID) continuous daily dosing in combination with Nivolumab administered intravenously (IV) at 3mg/kg Q2W
  Interventions: Drug: Nivolumab; Drug: Epacadostat
- Phase 1 Part 1 Epacadostat 50mg BID +Nivolumab (Experimental): Epacadostat 50mg oral twice daily (BID) continuous daily dosing in combination with Nivolumab administered intravenously (IV) at 3mg/kg Q2W
  Interventions: Drug: Nivolumab; Drug: Epacadostat
- Phase 1 Part 1 Epacadostat 100mg BID +Nivolumab (Experimental): Epacadostat 100mg oral twice daily (BID) continuous daily dosing in combination with Nivolumab administered intravenously (IV) at 3mg/kg Q2W.
  Interventions: Drug: Nivolumab; Drug: Epacadostat
- Phase 1 Part 1 Epacadostat 300mg BID +Nivolumab (Experimental): Epacadostat 300mg oral twice daily (BID) continuous daily dosing in combination with Nivolumab administered intravenously (IV) at 3mg/kg Q2W.
  Interventions: Drug: Nivolumab; Drug: Epacadostat
- Phase 1 Part 2 Epacadostat 100mg BID +Nivolumab +5-FU/Platinum (Experimental): Epacadostat 100mg oral twice daily (BID) continuous daily dosing in combination with Nivolumab 360mg Q3W and 5-FU/Platinum( Carboplatin or Cisplatin+5-Fluorouracil) administered intravenously (IV).
  Interventions: Drug: Nivolumab; Drug: Epacadostat; Drug: Chemotherapy
- Phase 1 Part 2 Epacadostat 100mg BID +Pemetrexed/Platinum (Experimental): Epacadostat 100mg oral twice daily (BID) continuous daily dosing in combination with Nivolumab 360 mg Q3W and Pemetrexed/Platinum (Carboplatin orCisplatin+Pemetrexed) administered intravenously (IV).
  Interventions: Drug: Epacadostat; Drug: Chemotherapy
- Phase 1 Part 2 Epacadostat 100mg BID +Paclitaxel/Platinum (Experimental): Epacadostat 100mg oral twice daily (BID) continuous daily dosing in combination with Nivolumab 360 mg Q3W and Paclitaxel/Platinum(Carboplatin+Cisplatin+Paclitaxel)administered intravenously (IV).
  Interventions: Drug: Epacadostat; Drug: Chemotherapy
- Phase 2 Epacadostat 100mg BID + Nivolumab (Experimental): Epacadostat 100mg oral twice daily (BID) continuous daily dosing in combination with Nivolumab 240mg Q2W or 480 mg Q4W based on tumor type administered intravenously (IV).
  Interventions: Drug: Nivolumab; Drug: Epacadostat
- Phase 2 Epacadostat 300mg BID + Nivolumab (Experimental): Epacadostat 300mg oral twice daily (BID) continuous daily dosing in combination with Nivolumab 240mg Q2W administered intravenously (IV).
  Interventions: Drug: Nivolumab; Drug: Epacadostat

INTERVENTIONS:
Drug: Nivolumab — specified dose and dosing schedule
  Arms: Phase 1 Part 1 Epacadostat 100mg BID +Nivolumab; Phase 1 Part 1 Epacadostat 25mg BID +Nivolumab; Phase 1 Part 1 Epacadostat 300mg BID +Nivolumab; Phase 1 Part 1 Epacadostat 50mg BID +Nivolumab; Phase 1 Part 2 Epacadostat 100mg BID +Nivolumab +5-FU/Platinum; Phase 2 Epacadostat 100mg BID + Nivolumab; Phase 2 Epacadostat 300mg BID + Nivolumab
Drug: Epacadostat — oral twice daily continuous at the protocol-defined dose
Drug: Chemotherapy — Specified dose on specified days
  Arms: Phase 1 Part 2 Epacadostat 100mg BID +Nivolumab +5-FU/Platinum; Phase 1 Part 2 Epacadostat 100mg BID +Paclitaxel/Platinum; Phase 1 Part 2 Epacadostat 100mg BID +Pemetrexed/Platinum

SUMMARY:
This is a Phase 1/2, open label study. Phase 1 consists of 2 parts. Part 1 is a dose-escalation assessment of the safety and tolerability of epacadostat administered with nivolumab in subjects with select advanced solid tumors and lymphomas. Part 2 will evaluate the safety and tolerability of epacadostat in combination with nivolumab and chemotherapy in subjects with squamous cell carcinoma of head and neck (SCCHN) and non-small cell lung cancer (NSCLC).

Phase 2 will include expansion cohorts in 7 tumor types, including melanoma, NSCLC, SCCHN, colorectal cancer, ovarian cancer, glioblastoma and diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age 18 years or older
* Subjects with histologically or cytologically confirmed NSCLC, MEL (including I/O relapsed MEL or I/O refractory MEL), CRC, SCCHN, ovarian cancer, recurrent B cell NHL or HL, or glioblastoma
* Presence of measurable disease by RECIST v1.1 for solid tumors or Cheson criteria for B cell NHL (including DLBCL) or HL. For subjects with glioblastoma, presence of measurable disease is not required.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Fresh baseline tumor biopsies (defined as a biopsy specimen taken since completion of the most recent prior chemotherapy regimen) are required for all cohorts except glioblastoma

Exclusion Criteria:

* Laboratory and medical history parameters not within Protocol-defined range
* Currently pregnant or breastfeeding
* Subjects who have received prior immune checkpoint inhibitors or an IDO inhibitor (except select Phase 2 cohorts evaluating I/O relapsed or I/O refractory MEL). Subjects who have received experimental vaccines or other immune therapies should be discussed with the medical monitor to confirm eligibility
* Untreated central nervous system (CNS) metastases or CNS metastases that have progressed
* Subjects with any active or inactive autoimmune process
* Evidence of interstitial lung disease or active, noninfectious pneumonitis
* Subjects with any active or inactive autoimmune process
* Ocular MEL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, Study Director — Incyte Corporation
Locations (24):
- United States (22):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - USC Norris Cancer Center, Los Angeles, California
  - UCSF - University of California San Francisco, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - NYU Cancer Center, New York, New York
  - Columbia University, Herbert Irving Comprehensive Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Medical Center Boulevard, Winston-Salem, North Carolina
  - Sanford Research, Fargo, North Dakota
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Sanford Research, North Sioux City, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology Research, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Trust, Oxford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 22 study sites in the United States and 2 study sites in the United Kingdom from 26 November 2014 to 16 June 2020.
Pre-assignment Details: A total of 307 participants were enrolled in this study, 48 participants were enrolled in Phase 1 and 259 participants were enrolled in Phase 2. Participants in Phase 1 Part 2 and Phase 2 received dose per select solid tumor types (Colorectal, Melanoma I/O Naïve, Melanoma I/O relapsed, Melanoma I/O refractory, Non-small cell lung cancer (NSCLC), Ovarian, Squamous cell carcinoma of the head and neck (SCCHN), Diffuse large B-cell lymphoma (DLBCL) and Glioblastoma).
Groups:
- Phase 1, Part 1: Epacadostat 25 mg + Nivolumab 3 mg: Participants received epacadostat 25 mg, orally, twice daily (BID) in combination of nivolumab 3 mg/kg intravenously (IV), on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 1, Part 1: Epacadostat 50 mg + Nivolumab 3 mg: Participants received epacadostat 50 mg, orally, BID in combination of nivolumab 3 mg/kg, IV, once every 3 weeks (Q3W), on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 1, Part 1: Epacadostat 100 mg + Nivolumab 3 mg: Participants received epacadostat 100 mg, orally, BID in combination of nivolumab 3 mg/kg, IV, Q3W, on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 1, Part 1: Epacadostat 300 mg + Nivolumab 3 mg: Participants received epacadostat 300 mg, orally, BID in combination of nivolumab 3 mg/kg, IV, Q3W, on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum: Participants with select solid tumor types received epacadostat 100 mg BID in combination with nivolumab 360 mg, IV, once every 2 weeks (Q2W), on Day 1 of each 21-day cycle along with 5-FU/Platinum chemotherapy regimen IV. Participants were de-escalated to epacadostat 50 mg BID if 100 mg was not tolerated.
- Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Pemetrexed/ Platinum: Participants with select solid tumor types received epacadostat 100 mg BID in combination with nivolumab 360 mg, IV, Q2W, on Day 1 of each 21-day cycle along with Pemetrexed /Platinum chemotherapy regimen IV. Participants were de-escalated to epacadostat 50 mg BID if 100 mg was not tolerated.
- Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Paclitaxel/ Platinum: Participants with select solid tumor types received epacadostat 100 mg BID in combination with nivolumab 360 mg, IV, Q2W, on Day 1 of each 21-day cycle along with Paclitaxel/Platinum chemotherapy regimen IV. Participants were de-escalated to epacadostat 50 mg BID if 100 mg was not tolerated.
- Phase 2: Epacadostat 100 mg + Nivolumab 240/480 mg: Participants with select solid tumor types received epacadostat 100 mg BID in combination with nivolumab 240 mg IV infusion Q2W on Days 1, 15, 29, and 43 and participants with melanoma I/O-relapsed and melanoma I/O-refractory enrolled in this arm received epacadostat 100 mg BID in combination with nivolumab 480 mg IV infusion once every 4 weeks (Q4W) on Days 1 and Day 29 of each 8-week cycle.
- Phase 2: Epacadostat 300 mg + Nivolumab 240 mg: Participants with select solid tumor types received epacadostat 300 mg BID in combination with nivolumab 240 mg IV infusion Q2W on Days 1, 15, 29, and 43 of each 8-week cycle.
Period: Overall Study
Arm/Group | Phase 1, Part 1: Epacadostat 25 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 50 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 100 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 300 mg + Nivolumab 3 mg | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Pemetrexed/ Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Paclitaxel/ Platinum | Phase 2: Epacadostat 100 mg + Nivolumab 240/480 mg | Phase 2: Epacadostat 300 mg + Nivolumab 240 mg
Started | 3 | 6 | 14 | 13 | 6 | 3 | 3 | 83 | 176
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 14 | 13 | 6 | 3 | 3 | 83 | 176
Not completed — Participants Decision: Consent Withdrawal from Study and Follow-up | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 11 | 25
Not completed — Death | 2 | 4 | 10 | 6 | 4 | 3 | 2 | 51 | 97
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 5
Not completed — Site Terminated by Sponsor | 1 | 0 | 1 | 4 | 0 | 0 | 0 | 11 | 25
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Completed 100 Day Safety Follow-up Period | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 11
Not completed — Reason not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 12

BASELINE CHARACTERISTICS:
Population: The safety population included all participants enrolled in the study who received at least 1 dose of epacadostat, nivolumab, or an applicable chemotherapy regimen.
Groups:
- Phase 1, Part 1: Epacadostat 25 mg + Nivolumab 3 mg: Participants received epacadostat 25 mg, orally, BID in combination of nivolumab 3 mg/kg, IV, on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 1, Part 1: Epacadostat 50 mg + Nivolumab 3 mg: Participants received epacadostat 50 mg, orally, BID in combination of nivolumab 3 mg/kg, IV, Q3W, on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum: Participants with select solid tumor types received epacadostat 100 mg BID in combination with nivolumab 360 mg, IV, Q2W, on Day 1 of each 21-day cycle along with 5-FU/Platinum chemotherapy regimen IV. Participants were de-escalated to epacadostat 50 mg BID if 100 mg was not tolerated.
- Phase 2: Epacadostat 100 mg + Nivolumab 240/480 mg: Participants with select solid tumor types received epacadostat 100 mg BID in combination with nivolumab 240 mg IV infusion Q2W on Days 1, 15, 29, and 43 and participants with melanoma I/O-relapsed and melanoma I/O-refractory enrolled in this arm received epacadostat 100 mg BID in combination with nivolumab 480 mg IV infusion Q4W on Days 1 and Day 29 of each 8-week cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 1, Part 1: Epacadostat 25 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 50 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 100 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 300 mg + Nivolumab 3 mg | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Pemetrexed/ Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Paclitaxel/ Platinum | Phase 2: Epacadostat 100 mg + Nivolumab 240/480 mg | Phase 2: Epacadostat 300 mg + Nivolumab 240 mg | Total
Number analyzed (Participants) | 3 | 6 | 14 | 13 | 6 | 3 | 3 | 83 | 176 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (26.00) | 62.5 (12.41) | 57.5 (13.27) | 61.6 (10.67) | 64.3 (6.38) | 67.7 (6.43) | 70.3 (11.37) | 56.7 (13.82) | 62.6 (12.12) | 60.7 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 11 | 5 | 1 | 1 | 1 | 46 | 77 | 145
  Male | 1 | 5 | 3 | 8 | 5 | 2 | 2 | 37 | 99 | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 11 | 17
  Not Hispanic or Latino | 3 | 5 | 14 | 13 | 6 | 3 | 3 | 77 | 159 | 283
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 4 | 7
  White | 3 | 6 | 13 | 13 | 5 | 3 | 3 | 76 | 160 | 282
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Phase 1, Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as occurrence of any treatment-emergent adverse event (TEAE) in Phase 1 Parts 1 and 2. DLT included all TEAE of specified grades such as 1) Hematologic toxicities - any Grade 4 thrombocytopenia or neutropenia, anemia, febrile neutropenia, ≥ Grade 3 hemolysis, thrombocytopenia and 2) Nonhematologic toxicities - Grade 4 AE, nausea, vomiting, or diarrhea, electrolyte abnormality, ≥ Grade 3 aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin elevation, Grade 2 AST/ALT with symptomatic liver inflammation, AST or ALT > 3 × upper limit of normal (ULN) and concurrent total bilirubin > 2 × ULN without initial findings of cholestasis, and any other ≥ Grade 3 toxicity. A TEAE is any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and up to 100 days after last dose of study drug.
Time Frame: Day 42
Population: The Phase 1, Part 1 Safety Population includes all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Part 1: Epacadostat 25 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 50 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 100 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 300 mg + Nivolumab 3 mg
Number analyzed (Participants) | 3 | 6 | 14 | 13
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1, Part 2: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: as for outcome 1
Time Frame: Day 42
Population: The Phase 1, Part 2 Safety Population includes all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Pemetrexed/ Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Paclitaxel/ Platinum
Number analyzed (Participants) | 6 | 3 | 3
Participants | 0 | 0 | 0

3. Primary Outcome: Phase 1, Parts 1 and 2: Number of Participants With At Least One Treatment-Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and up to 100 days after last dose of study drug.
Time Frame: up to approximately 39 months
Population: The Phase 1, Parts 1 and 2 Safety Population includes all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Part 1: Epacadostat 25 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 50 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 100 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 300 mg + Nivolumab 3 mg | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Pemetrexed/ Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Paclitaxel/ Platinum
Number analyzed (Participants) | 3 | 6 | 14 | 13 | 6 | 3 | 3
Participants | 3 | 6 | 14 | 13 | 6 | 3 | 3

4. Primary Outcome: Phase 2: Objective Response Rate (ORR) in Participants With Select Solid Tumors Per Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 for Participants With Solid Tumors and Per Cheson Criteria for Participants With DLBCL
Description: ORR was defined as the percentage of participants having a complete response (CR) or partial response (PR) as determined by investigator assessment of radiographic disease per RECIST v1.1. CR per RECIST v 1.1 was defined as disappearance of all target lesions. PR per RECIST v 1.1 was defined as At least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the Baseline sum diameters. Data is reported as per dose received by the participants with a particular cancer type. CR per Cheson criteria was defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms. PR per Cheson criteria was defined as at least a 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses.
Time Frame: From first dose up end of the study (up to approximately 6 years)
Population: The Phase 2 Full Analysis Population includes all participants enrolled in the study who received at least 1 dose of study drug. The data is reported per cancer type in this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Phase 2: Epacadostat 100 mg + Nivolumab 240 in Colorectal Cancer: Participants with Colorectal Cancer received epacadostat 100 mg BID in combination with nivolumab 240 mg IV infusion Q2W on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 2: Epacadostat 300 mg + Nivolumab 240 mg in DLBCL: Participants with DLBCL received epacadostat 300 mg BID in combination with nivolumab 240 mg IV infusion Q2W on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 2: Epacadostat 100/300 mg + Nivolumab 240 mg in Melanoma(I/O Naive): Participants with Melanoma(I/O Naive) received epacadostat 100 mg or 300 mg BID in combination with nivolumab 240 mg IV infusion Q2W on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 2 Epacadostat 100mg + Nivolumab 480 mg in Melanoma (I/O Relapsed): Participants with Melanoma (I/O Relapsed) received epacadostat 100 mg BID in combination with nivolumab 480 mg IV infusion Q2W on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 2 Epacadostat 100mg + Nivolumab 480 mg in Melanoma (I/O Refractory): Participants with Melanoma (I/O Refractory) received epacadostat 100 mg BID in combination with nivolumab 480 mg IV infusion Q2W on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in NSCLC: Participants with NSCLC received epacadostat 100 mg or 300 mg BID in combination with nivolumab 240 mg IV infusion Q2W on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in Ovarian Cancer: Participants with Ovarian Cancer received epacadostat 100 mg or 300 mg BID in combination with nivolumab 240 mg IV infusion Q2W on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in SCCHN: Participants with SCCHN received epacadostat 100/300 mg BID in combination with nivolumab 240 mg IV infusion Q2W on Days 1, 15, 29, and 43 of each 8-week cycle.
- Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in Glioblastoma: Participants with Glioblastoma received epacadostat 100/300 mg BID in combination with nivolumab 240 mg IV infusion Q2W on Days 1, 15, 29, and 43 of each 8-week cycle.
Arm/Group | Phase 2: Epacadostat 100 mg + Nivolumab 240 in Colorectal Cancer | Phase 2: Epacadostat 300 mg + Nivolumab 240 mg in DLBCL | Phase 2: Epacadostat 100/300 mg + Nivolumab 240 mg in Melanoma(I/O Naive) | Phase 2 Epacadostat 100mg + Nivolumab 480 mg in Melanoma (I/O Relapsed) | Phase 2 Epacadostat 100mg + Nivolumab 480 mg in Melanoma (I/O Refractory) | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in NSCLC | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in Ovarian Cancer | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in SCCHN | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in Glioblastoma
Number analyzed (Participants) | 26 | 18 | 50 | 7 | 7 | 58 | 29 | 31 | 33
percentage of participants | 3.8 | 0.0 | 62.0 | 28.6 | 28.6 | 20.7 | 13.8 | 25.8 | 0.0

5. Primary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first documented progressive disease per RECIST v1.1 or death due to any cause, whichever occurs first.
Time Frame: From first dose up end of the study (up to approximately 6 years)
Population: The Phase 2 Full Analysis Population includes all participants enrolled in the study who take at least 1 dose of study drug. The data is reported per cancer type in this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Epacadostat 100 mg + Nivolumab 240 in Colorectal Cancer | Phase 2: Epacadostat 300 mg + Nivolumab 240 mg in DLBCL | Phase 2: Epacadostat 100/300 mg + Nivolumab 240 mg in Melanoma(I/O Naive) | Phase 2 Epacadostat 100mg + Nivolumab 480 mg in Melanoma (I/O Relapsed) | Phase 2 Epacadostat 100mg + Nivolumab 480 mg in Melanoma (I/O Refractory) | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in NSCLC | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in Ovarian Cancer | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in SCCHN | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in Glioblastoma
Number analyzed (Participants) | 26 | 18 | 50 | 7 | 7 | 58 | 29 | 31 | 33
months | 1.78 [1.74 to 1.81] | 1.64 [1.35 to 3.52] | NA [9.51 to NA] — Median and upper limit of 95% confidence interval (CI) was not estimable due to low number of participants with events. | 1.76 [0.46 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 2.55 [0.59 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 1.88 [1.78 to 2.04] | 1.88 [1.68 to 3.52] | 3.62 [1.78 to 9.08] | 1.84 [1.78 to 2.63]

6. Primary Outcome: Phase 2: Overall Survival (OS) Rate of Proportion With Glioblastoma
Description: OS rate is defined as the proportion of participants alive 9 months after the start of treatment.
Time Frame: Month 9
Population: The Phase 2 Full Analysis Population includes all participants enrolled in the study who take at least 1 dose of study drug. The data is reported for participants with Glioblastoma cancer type for this outcome measure.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Phase 2: Epacadostat 100/300 mg + Nivolumab 240 mg: Participants with Glioblastoma received epacadostat 100/300 mg BID in combination with nivolumab 240 mg IV infusion Q2W on Days 1, 15, 29, and 43 of each 8-week cycle.
Arm/Group | Phase 2: Epacadostat 100/300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 33
proportion of participants | 0.458 [0.297 to 0.605]

7. Secondary Outcome: Phase 1, Part 2: ORR Per RECIST v1.1 and for Participants With Advanced or Metastatic SCCHN and Advanced or Metastatic NSCLC
Description: ORR was defined as percentage of participants having CR or PR as determined by investigator assessment of radiographic disease per RECIST v1.1. CR per RECIST v 1.1 was defined as disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the Baseline sum diameters.
Time Frame: From first dose up end of the study (up to approximately 6 years)
Population: The Phase 1, Part 2 Full Analysis Population includes all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Pemetrexed/ Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Paclitaxel/ Platinum
Number analyzed (Participants) | 6 | 3 | 3
percentage of participants | 50.0 | 33.3 | 100.0

8. Secondary Outcome: Phase 1, Part 1: ORR Per RECIST v1.1 for Participants With Solid Tumors; Per Cheson Criteria for Participants With B-cell NHL; and Per RANO and mRANO Criteria for Participants With GBM
Description: ORR was defined as percentage of participants having CR or PR as determined by investigator assessment of radiographic disease per RECIST v1.1. CR per RECIST v 1.1 was defined as disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the Baseline sum diameters. Per Cheson criteria, CR: complete disappearance of all detectable clinical evidence of disease and disease-related symptoms. PR: at least a 50% decrease in SPD of up to 6 of the largest dominant nodes or nodal masses. Per RANO criteria, CR: Complete disappearance of all enhancing measurable and non-measurable disease sustained. PR: at least ≥50% decrease compared with baseline in the SOD of all measurable enhancing lesions sustained.
Time Frame: From first dose up end of the study (up to approximately 6 years)
Population: The Phase 1, Part 1 Full Analysis Population includes all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1, Part 1: Epacadostat 25 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 50 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 100 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 300 mg + Nivolumab 3 mg
Number analyzed (Participants) | 3 | 6 | 14 | 13
percentage of participants | 0.0 | 0.0 | 0.0 | 23.1

9. Secondary Outcome: Phase 1, Part 2: Duration of Response (DOR) for Participants With Advanced or Metastatic SCCHN and Advanced or Metastatic NSCLC
Description: DOR is defined as the time from the first overall response contributing to an objective response (CR or PR) to the earlier of the participant's death and first overall response of PD. CR was defined as disappearance of all target lesions. PR was defined as At least a 30% decrease in the SOD of target lesions, taking as reference the Baseline sum diameters. PD was defined as at least a 20% increase in the SOD of target lesions.
Time Frame: From first dose up end of the study (up to approximately 6 years)
Population: The Phase 1, Part 2 Full Analysis Population includes all participants enrolled in the study who received at least 1 dose of study drug. The data is reported only for responders for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Pemetrexed/ Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Paclitaxel/ Platinum
Number analyzed (Participants) | 3 | 1 | 3
months | 3.82 [3.75 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median value can't be reported for a single participant due to the risk of patient re-identification. | 3.93 [2.76 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died.

10. Secondary Outcome: Phase 1, Part 2: PFS for Participants With Advanced or Metastatic SCCHN and Advanced or Metastatic NSCLC
Description: PFS is defined as the time from randomization to the first documented progressive disease or death due to any cause, whichever occurs first.
Time Frame: From first dose up end of the study (up to approximately 6 years)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Pemetrexed/ Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Paclitaxel/ Platinum
Number analyzed (Participants) | 6 | 3 | 3
months | 5.72 [2.07 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 2.83 [1.35 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 6.10 [4.84 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died.

11. Secondary Outcome: Phase 2: Duration of Response
Description: DOR is defined as the time from the first overall response contributing to an objective response (CR or PR) to the earlier of the participant's death and first overall response of PD. CR was defined as disappearance of all target lesions. PR was defined as At least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the Baseline sum diameters. PD was defined as at least a 20% increase in the SOD of target lesions.
Time Frame: From first dose up end of the study (up to approximately 6 years)
Population: The Phase 2 Full Analysis Population includes all participants enrolled in the study who received at least 1 dose of study drug. The data is reported only for responders and per cancer type for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Epacadostat 100 mg + Nivolumab 240 in Colorectal Cancer | Phase 2: Epacadostat 300 mg + Nivolumab 240 mg in DLBCL | Phase 2: Epacadostat 100/300 mg + Nivolumab 240 mg in Melanoma(I/O Naive) | Phase 2 Epacadostat 100mg + Nivolumab 480 mg in Melanoma (I/O Relapsed) | Phase 2 Epacadostat 100mg + Nivolumab 480 mg in Melanoma (I/O Refractory) | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in NSCLC | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in Ovarian Cancer | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in SCCHN | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in Glioblastoma
Number analyzed (Participants) | 1 | 0 | 31 | 1 | 2 | 12 | 4 | 8 | 0
months | NA [NA to NA] — Median, lower and upper limit of 95% CI was not estimable for 1 participant. |  | NA [NA to NA] — Median, lower and upper limit of 95% CI was not estimable due to low number of participants with events. | NA [NA to NA] — Median, lower and upper limit of 95% CI was not estimable for 1 participant. | NA [NA to NA] — Median and 95% CI was not estimable due to low number of participants with events. | NA [1.94 to NA] — Median and upper limit of 95% CI was not estimable due to low number of participants with events. | 3.93 [3.13 to 5.53] | NA [7.37 to NA] — Median and upper limit of 95% CI was not estimable due to low number of participants with events. |

12. Secondary Outcome: Phase 2: Duration of Disease Control, Defined as CR, PR, and Stable Disease (SD)
Description: Duration of disease control is the time from the first dose to the first objective response of PD, or death, whichever occurs first, for participants who reported a best overall response of SD or better. PD was defined as at least a 20% increase in the SOD of target lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the Baseline sum diameters.
Time Frame: From first dose up end of the study (up to approximately 6 years)
Population: The Phase 2 Full Analysis Population includes all participants enrolled in the study who received at least 1 dose of study drug. The data is reported per cancer type in this outcome measure. Overall number analyzed are the participants who had best overall response of stable disease or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Epacadostat 100 mg + Nivolumab 240 in Colorectal Cancer | Phase 2: Epacadostat 300 mg + Nivolumab 240 mg in DLBCL | Phase 2: Epacadostat 100/300 mg + Nivolumab 240 mg in Melanoma(I/O Naive) | Phase 2 Epacadostat 100mg + Nivolumab 480 mg in Melanoma (I/O Relapsed) | Phase 2 Epacadostat 100mg + Nivolumab 480 mg in Melanoma (I/O Refractory) | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in NSCLC | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in Ovarian Cancer | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in SCCHN | Phase 2 Epacadostat 100/300 mg + Nivolumab 240 mg in Glioblastoma
Number analyzed (Participants) | 4 | 4 | 39 | 2 | 3 | 19 | 9 | 17 | 8
months | 3.72 [2.86 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 4.57 [3.52 to 10.26] | NA [NA to NA] — Median, lower and upper limit of 95% CI was not estimable due to low number of participants with events. | NA [NA to NA] — Median, lower and upper limit of 95% CI was not estimable due to low number of participants with events. | NA [3.19 to NA] — Median, and upper limit of 95% CI was not estimable due to low number of participants with events. | NA [9.11 to NA] — Median, and upper limit of 95% CI was not estimable due to low number of participants with events. | 5.86 [3.52 to 7.47] | 10.89 [4.84 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 3.72 [3.49 to 5.59]

13. Secondary Outcome: Phase 2: Safety and Tolerability Measured by the Number of Adverse Events (AEs), Serious Adverse Events (SAEs), and Fatal Treatment Emergent AEs
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and up to 100 days after last dose of study drug. Adverse events of grade 5 which result in death are called as fatal AEs.
Time Frame: up to approximately 35 months
Population: The Phase 2 Safety population includes all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Epacadostat 100 mg + Nivolumab 240/480 mg | Phase 2: Epacadostat 300 mg + Nivolumab 240 mg
Number analyzed (Participants) | 83 | 176
Participants
  Participants with Treatment Emergent Adverse Events | 82 | 176
  Participants with Serious Treatment Emergent AEs | 40 | 89
  Participants with Fatal Treatment Emergent AEs | 4 | 5

ADVERSE EVENTS:
Time Frame: up to approximately 39 months for Phase 1 and up to approximately 35 months for Phase 2
Description: The safety population includes all subjects enrolled in the study who received at least 1 dose of study drug .
Groups:
- Total: Total
Arm/Group | Phase 1, Part 1: Epacadostat 25 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 50 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 100 mg + Nivolumab 3 mg | Phase 1, Part 1: Epacadostat 300 mg + Nivolumab 3 mg | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Pemetrexed/ Platinum | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Paclitaxel/ Platinum | Phase 2: Epacadostat 100 mg + Nivolumab 240/480 mg | Phase 2: Epacadostat 300 mg + Nivolumab 240 mg | Total
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/6 | 11/14 | 7/13 | 4/6 | 3/3 | 2/3 | 52/83 | 97/176 | 182/307
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/6 | 4/14 | 4/13 | 4/6 | 2/3 | 2/3 | 40/83 | 89/176 | 148/307
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 14/14 | 13/13 | 6/6 | 3/3 | 3/3 | 81/83 | 173/176 | 302/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Part 1: Epacadostat 25 mg + Nivolumab 3 mg (N=3) | Phase 1, Part 1: Epacadostat 50 mg + Nivolumab 3 mg (N=6) | Phase 1, Part 1: Epacadostat 100 mg + Nivolumab 3 mg (N=14) | Phase 1, Part 1: Epacadostat 300 mg + Nivolumab 3 mg (N=13) | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum (N=6) | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Pemetrexed/ Platinum (N=3) | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Paclitaxel/ Platinum (N=3) | Phase 2: Epacadostat 100 mg + Nivolumab 240/480 mg (N=83) | Phase 2: Epacadostat 300 mg + Nivolumab 240 mg (N=176) | Total (N=307)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Adrenocortical insufficiency acute (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Central nervous system infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 6 (6) | 11 (12)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 7 (8)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Exsanguination (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Hemianopia homonymous (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 4 (4) | 9 (10)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 6 (6)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 5 (7)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (7) | 7 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (6) | 7 (8)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 8 (9) | 15 (17)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 6 (7)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 5 (6)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 6 (6)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 7 (9)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (8) | 8 (10)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Part 1: Epacadostat 25 mg + Nivolumab 3 mg (N=3) | Phase 1, Part 1: Epacadostat 50 mg + Nivolumab 3 mg (N=6) | Phase 1, Part 1: Epacadostat 100 mg + Nivolumab 3 mg (N=14) | Phase 1, Part 1: Epacadostat 300 mg + Nivolumab 3 mg (N=13) | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + 5-FU/Platinum (N=6) | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Pemetrexed/ Platinum (N=3) | Phase 1, Part 2: Epacadostat 100 mg + Nivolumab 360 mg + Paclitaxel/ Platinum (N=3) | Phase 2: Epacadostat 100 mg + Nivolumab 240/480 mg (N=83) | Phase 2: Epacadostat 300 mg + Nivolumab 240 mg (N=176) | Total (N=307)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 13 (13)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 14 (19) | 18 (20) | 43 (50)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 7 (7) | 12 (12)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 12 (17) | 37 (51) | 53 (73)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 8 (9)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 9 (15) | 16 (21) | 29 (43)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 4 (4) | 1 (2) | 2 (2) | 17 (22) | 30 (42) | 62 (80)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 12 (12) | 19 (20)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 12 (13) | 25 (33) | 42 (54)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 17 (27) | 39 (58) | 61 (93)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 11 (12) | 30 (35) | 45 (51)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 7 (7)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 15 (25) | 23 (27) | 40 (54)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 4 (4) | 9 (12)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 16 (26) | 13 (21) | 35 (53)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 4 (6)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 5 (7)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Carcinoembryonic antigen increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 10 (11) | 8 (10) | 22 (25)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 7 (10) | 11 (14)
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (2) | 2 (3) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 25 (26) | 51 (57) | 90 (99)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 7 (7)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 3 (5)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 2 (3) | 19 (23) | 41 (50) | 72 (86)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 7 (7) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 22 (24) | 62 (69) | 98 (109)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 19 (28) | 25 (34)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 11 (11) | 18 (18)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (9) | 9 (11)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (7) | 1 (1) | 3 (5) | 2 (4) | 4 (6) | 1 (3) | 0 (0) | 25 (32) | 58 (91) | 96 (149)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (13) | 28 (32) | 42 (49)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 9 (9)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 7 (7) | 10 (11) | 19 (20)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 10 (10)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 3 (3) | 14 (14) | 24 (25)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 13 (13) | 24 (24)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 8 (8) | 14 (15)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 1 (4) | 1 (1) | 0 (0) | 21 (22) | 30 (34) | 59 (68)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 8 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 6 (8)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 8 (8)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 21 (24) | 28 (31)
Fatigue (General disorders) | 3 (3) | 3 (3) | 4 (4) | 2 (3) | 4 (6) | 3 (4) | 2 (2) | 36 (38) | 123 (131) | 180 (194)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 7 (7)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 9 (9) | 16 (16)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 6 (6)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 0 (0) | 8 (10)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 2 (4) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 15 (17) | 40 (52) | 64 (80)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (12) | 11 (14)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 4 (4) | 8 (9)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 6 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (10) | 12 (17) | 21 (28)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 13 (17) | 16 (32) | 31 (51)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 8 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (14) | 3 (8) | 12 (24)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 7 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 14 (16) | 21 (24)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 9 (13) | 14 (18)
Hypogonadism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 12 (20) | 14 (18) | 33 (46)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 7 (12) | 14 (23)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 13 (23) | 28 (35) | 45 (62)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 10 (16) | 14 (21)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (7) | 16 (18) | 23 (26)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 12 (13) | 20 (21) | 37 (39)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 9 (10) | 15 (17)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (4) | 7 (9)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 8 (10) | 15 (19)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 9 (9) | 25 (25) | 43 (43)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 4 (12) | 1 (1) | 0 (0) | 0 (0) | 8 (11) | 20 (28) | 35 (55)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (12) | 14 (18) | 20 (30)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (5)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 10 (11)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 6 (6) | 10 (10)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 6 (6) | 12 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 13 (13) | 18 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 12 (12) | 10 (13) | 29 (34)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 20 (24) | 26 (30)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 7 (9)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 6 (6) | 3 (3) | 3 (6) | 0 (0) | 2 (2) | 30 (35) | 75 (99) | 122 (155)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 8 (8) | 18 (18)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (7) | 10 (10)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 6 (7)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 9 (9) | 11 (11)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 15 (18) | 17 (18) | 37 (41)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 13 (16) | 19 (25)
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 11 (13) | 17 (19)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Pancreatic insufficiency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 11 (13) | 15 (17)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 5 (5) | 12 (12)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (14) | 5 (5) | 13 (22)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 8 (8)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 12 (12)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 4 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 6 (6)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 7 (7)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 10 (11) | 12 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 1 (1) | 4 (4) | 4 (5) | 0 (0) | 0 (0) | 16 (27) | 34 (44) | 62 (86)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 7 (8)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 12 (16) | 29 (41) | 48 (66)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 5 (7) | 4 (4) | 0 (0) | 0 (0) | 1 (2) | 19 (25) | 39 (50) | 69 (89)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 5 (7)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 11 (14) | 29 (32) | 43 (49)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 3 (3) | 8 (11)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 6 (6)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 4 (5) | 9 (10)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 6 (6)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 10 (10) | 15 (17)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 6 (7) | 13 (17)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (9) | 0 (0) | 0 (0) | 5 (5) | 14 (15) | 25 (30)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Suprapubic pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 6 (8) | 16 (18)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Tracheal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 6 (6) | 11 (11)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 13 (20) | 24 (33)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 8 (8)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (4) | 1 (1) | 0 (0) | 6 (14) | 13 (20) | 25 (43)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 5 (6)
Vaginal odour (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 4 (4) | 9 (10) | 18 (20)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 3 (3) | 6 (9)
Vitamin B1 decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (6) | 2 (5) | 0 (0) | 1 (1) | 17 (21) | 43 (64) | 71 (101)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 9 (9) | 26 (29) | 44 (47)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 5 (5) | 12 (14)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 7 (9) | 11 (13)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 9 (12) | 13 (16)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT02327078/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT02327078/SAP_001.pdf